CLINICAL TRIAL: NCT05528380
Title: Development of a Lifestyle Physical Activity Intervention to Reduce Risk for Perinatal Cannabis Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA055317-01A1 (NIH)
Record Dates: First submitted 2022-07-19; First posted 2022-09-06 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Pregnancy; Cannabis
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCT Intervention (Experimental): In the Open Trial all participants received a Fitbit to track activity levels and participate in a 6-session lifestyle physical activity intervention over the course of 12 weeks. The intervention consists of 20-25 minute phone or video-delivered session to: (a) review PA progress and re-evaluate current step-count goals, (b) problem-solve barriers to incorporating PA into their daily lives, (c) address difficulties utilizing the Fitbit, (d) encourage the use of bouts of PA as a coping strategy, and e) engage the participant in brief discussions focused on increasing and maintaining PA.
  Interventions: Behavioral: LPA + Fitbit Intervention
- Fitbit Only (Active Comparator): Participants randomly assigned to this are will receive a Fitbit to track activity levels and participate in 6 brief check-ins to assess any issues with the Fitbit device or app.
  Interventions: Behavioral: Fitbit Only

INTERVENTIONS:
Behavioral: LPA + Fitbit Intervention — Participants will receive a Fitbit to track activity levels and participate in a 6-session lifestyle physical activity intervention over the course of 12 weeks. The intervention consists of 20-25 minute phone or video-delivered session to: (a) review PA progress and re-evaluate current step-count goals, (b) problem-solve barriers to incorporating PA into their daily lives, (c) address difficulties utilizing the Fitbit, (d) encourage the use of bouts of PA as a coping strategy, and e) engage the participant in brief discussions focused on increasing and maintaining PA.
  Other Names: Women Out Walking
  Arms: RCT Intervention
Behavioral: Fitbit Only — Participants will receive a Fitbit to track activity levels and participate in 6 brief check-ins to assess any issues with the Fitbit device or app.
  Arms: Fitbit Only

SUMMARY:
This study will recruit 20 women who are high risk for prenatal cannabis use for a 12-week program of using the tracker and receiving a Lifestyle Physical Activity program. The primary outcomes will be self reported percent days of cannabis use and physical activity. Secondary outcomes include self -reported measures of depression and anxiety symptoms, adaptive coping, and self-efficacy for cannabis abstinence.

DETAILED DESCRIPTION:
This study will recruit 20 women in an open trial who are high risk for prenatal cannabis use for a 12-week program of using a Fitbit activity tracker and receiving a Lifestyle Physical Activity program. The primary outcomes will be self reported percent days of cannabis use and physical activity. Secondary outcomes include self -reported measures of depression and anxiety symptoms, adaptive coping, and self-efficacy for cannabis abstinence. The investigators will clinically monitor all participants in the study for safety and clinical deterioration, and measure a variety of symptom outcomes over the course of the intervention period during pregnancy, as well as at a postpartum follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18+
* 12-25 weeks gestation with a healthy singleton pregnancy
* Medically cleared for moderate physical activity
* Self-report of cannabis use at least once/week in the 3 months prior to the pregnancy desire to not engage in prenatal cannabis use
* Elevated depression (EPDS>=7) or anxiety (GAD7>=5)
* English-speaking
* Owns a smartphone to enable use of the Fitbit app
* Current physical activity does not meet health recommendations (150 min/week mod intensity activity)
* Expresses interest in reducing or discontinuing cannabis use

Exclusion Criteria:

* Current DSM-5 diagnosis of moderate/severe substance use disorder other than CUD or nicotine use disorder
* Use of illicit substances in the last 3 months (other than cannabis)
* Acute psychotic symptoms
* Current or recent suicidality or homicidally
* Current anorexia or bulimia
* Cognitive impairment
* Physical or medical problems that would not allow safe participation in moderate intensity PA (i.e., not medical cleared by Ob/Gyn)
* Has a plan to relocate away from the area during study period
* Recently started new mental health or substance use treatment within past 4 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-back (TLFB) | Baseline to 12-week endpoint
  Interviewer-administered assessment of use of cannabis, alcohol, tobacco, and other drugs
Steps/day | Baseline to 12-week endpoint
  objectively-measured
Activity Minutes/Day | Baseline to 12-week endpoint
  objectively-measured
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 1 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire -factor 1: daily sessions
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 2 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 2: frequency
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 3 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 3: age of onset
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 4 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 4: Marijuana quantity
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 5 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 5: Concentrate quantity
The Daily Sessions, Frequency & Quantity of Cannabis Use Inventory - Factor 6 | Baseline to 12-week endpoint
  Self-reported cannabis use questionnaire - factor 6: Edibles quantity
Urine Toxicology Screen | Baseline to 12-week endpoint
  Objective screening for use of cannabis via measurement of THC in urine samples
International Physical Activity Questionnaire | Baseline to 12-week endpoint
  self-report measure of physical activity including minutes/week spent walking, engaging in moderate physical activity, and engaging in vigorous physical activity

SECONDARY OUTCOMES:
Brief COPE | Baseline to 12-week endpoint
  Self-report measure of of use of coping strategies; includes 14 2-item scales, each ranging form 2-8. Higher scores indicate increased utilization of a coping strategy.
Marijuana Self-Efficacy Questionnaire | Baseline to 12-week endpoint
  Self-report measure of efficacy for cannabis abstinence; Scores range from 0-100, with higher scores indicating greater use of strategies to reduce marijuana consumption.
Edinburgh Postnatal Depression Screen | Baseline to 12-week endpoint
  Self-report measure of depression severity; scores range from 0-30, with higher scores indicating higher depression
Generalized Anxiety Disorder -7 | Baseline to 12-week endpoint
  Self-report measure of anxiety severity; scores range from 0-21, with higher scoring indicating more anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States